CLINICAL TRIAL: NCT04223531
Title: The Natriuretic Peptide Response to Saline Infusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Deepak Gupta, Assistant Professor of Medicine, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 191254
Record Dates: First submitted 2019-08-16; First posted 2020-01-10 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Saline (Other): Each participant will receive a saline infusion of normal saline 0.9%NaCl
  Interventions: Drug: Normal Saline 0.9% Infusion Solution Bag

INTERVENTIONS:
Drug: Normal Saline 0.9% Infusion Solution Bag — Participants will receive a normal saline infusion at a rate of 10ml per unit of body surface area per minute for 120 minutes.

SUMMARY:
The primary objective is to evaluate the overarching hypothesis that obese and black individuals have relatively lower circulating natriuretic peptide levels compared with lean and white individuals. Conventional clinical assays for measurement of circulating natriuretic peptides display substantial overlap, precluding determination of the basis of the relative natriuretic peptide deficiency previously observed in these groups. We will study lean or obese, black or white, healthy adult subjects with intravenous (IV) saline infusion as a stimulus for natriuretic peptide production and release. We will measure circulating levels of natriuretic peptide isoforms using mass spectrometry that allows the specific identification of proBNP 1-108 and its cleavage product BNP 1-32.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years;
* BMI between 18 and 25 (lean) or 30 and 40 kg/m2 (obese);
* self-reported race of either black or white;
* otherwise healthy with no chronic comorbidities.

Exclusion Criteria:

* History of diabetes mellitus
* Currently pregnant
* History of cardiac disorder including heart failure, cardiomyopathy, myocardial infarction, coronary revascularization, abnormal stress test, uncontrolled arrhythmia or arrhythmia requiring treatment, congenital heart disease, pericardial disease.
* History of hypertension defined as taking anti-hypertensive medications or untreated hypertension with systolic blood pressure ≥ 140 mm Hg or diastolic blood pressure ≥ 90 mm Hg at most recent clinical visit or screening visit.
* Obstructive lung disease
* History of chronic kidney disease
* History of liver disease or cirrhosis
* Uncontrolled thyroid dysfunction
* History of solid organ transplant
* History of malignancy other than basal or squamous cell skin cancer
* Inability to lie flat for 6 hours

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-06-17 (Actual)

PRIMARY OUTCOMES:
Change in circulating levels of proBNP 1-108 from baseline to 6 hours | Saline infusion will be given for 2 hours (with 4 hour observation) with blood samples collected at hourly intervals for 7 hours total
  proBNP 1-108 is a protein made by the heart. The change in circulating levels will be measured in response to saline infusion
Change in circulating levels of proBNP 1-32 from baseline to 6 hours | Saline infusion will be given for 2 hours (with 4 hour observation) with blood samples collected at hourly intervals for 7 hours total
  BNP 1-32 is a hormone made by the heart. The change in circulating levels will be measured in response to saline infusion

CONTACTS AND LOCATIONS:
Overall Officials: Deepak K Gupta, MD, MSCI, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Univeristy, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Only deidentified individual participant data will be provided to interested researchers with a data use agreement and confirmation that no protected health information will be shared, all data will be stored in password protected databases accessible to only key study personnel, and that data will be returned or destroyed after completion or 6 years, whichever is shorter.
Supporting Information: Study Protocol, SAP
Time Frame: No later than 1 year after completion of the study.
Access Criteria: Only deidentified individual participant data will be provided to interested researchers with a data use agreement and confirmation that no protected health information will be shared, all data will be stored in password protected databases accessible to only key study personnel, and that data will be returned or destroyed after completion or 6 years, whichever is shorter.